CLINICAL TRIAL: NCT03702192
Title: EXCOR® Pediatric VAD Anticoagulation IDE Investigational Plan
Brief Title: EXCOR® Pediatric VAD Anticoagulation IDE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI withdrew protocol
Sponsor: David N. Rosenthal (Other)
Responsible Party: Sponsor-Investigator, David N. Rosenthal, Professor of Pediatrics, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-47736
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Pediatric HD
Keywords: heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- single-arm novel anticoagulation (Experimental): Single-arm clinical study to assess the safety, and effectiveness of a novel anticoagulation protocol to be used in conjunction with the Berlin Heart EXCOR Pediatric Ventricular Assist Device as a bridge to heart transplantation in children with severe heart failure who have failed optimal medical therapy.
  Interventions: Device: novel anticoagulation protocol used in conjunction with the Berlin Heart EXCOR

INTERVENTIONS:
Device: novel anticoagulation protocol used in conjunction with the Berlin Heart EXCOR — novel antithrombotic management protocol

SUMMARY:
The Berlin Heart EXCOR ventricular assist device received approval from the FDA as a bridge to transplantation for children in 2011. Successful bridge to transplantation or recovery in the IDE trial of the Berlin Heart EXCOR was 88% to 92%, but a high incidence of neurological injury was reported in this trial (29%).

Stroke remains the most important complication of Berlin Heart EXCOR support, with high mortality rates, and considerable long-term morbidity. The EXCOR IDE study incorporated a novel anticoagulation protocol (henceforth referred to as the Edmonton Anticoagulation Protocol). The preponderance of ischemic strokes in this study raised the question of whether the anticoagulation protocol was sufficiently intensive, as ischemic strokes in this setting are virtually always thromboembolic phenomena. In response to these data and to the experience at the investigator's institution, a novel anticoagulation protocol has been devised for use with the EXCOR (Stanford anticoagulation protocol).The purpose of this study is to perform a pilot evaluation of this protocol in a multi--center setting, to prepare for a randomized trial between this and a subsequent iteration of anticoagulation treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Severe heart failure (NYHA functional class IV, or Ross functional class IV if < age 6 years of age), refractory to optimal medical therapy
2. Patient deemed to be candidate for EXCOR implantation according to the clinical criteria employed by treating site
3. Listed or eligible for cardiac transplantation according to the criteria employed by the treating site
4. Two-ventricle circulation, including cardiomyopathy, repaired structural heart disease, or acquired heart disease
5. Age 0 to 18 years of age
6. Corrected gestational age ≥ 37 weeks
7. Weight ≥ 3 kg and ≤ 60 kg
8. Legal guardian (and patient if age-appropriate) understands the nature of the investigation, is willing to comply with the protocol and associated evaluations, and provides written informed consent and assent prior to the procedure.

   -

Exclusion Criteria:

1. Support on ECMO for ≥10 days
2. Cardiopulmonary resuscitation (CPR) duration ≥ 30 minutes within 48 hours prior to device implantation
3. Body weight < 3.0 kg or BSA > 1.5 m2
4. Presence of mechanical aortic valve
5. Unfavorable or technically-challenging cardiac anatomy including single ventricle lesions, complex heterotaxy, and restrictive cardiomyopathy.
6. Evidence of intrinsic hepatic disease as defined by a total bilirubin level or ALT greater than 5 times the upper limit of normal for age, except in association with acute heart failure as determined by the site principal investigator
7. Evidence of intrinsic renal disease as defined by a serum creatinine greater than 3 times the upper limit of normal for age, except in association with acute heart failure as determined by the investigator
8. Hemodialysis or peritoneal dialysis (not including dialysis or continuous veno-venous hemofiltration (CVVH) for volume removal)
9. Evidence of intrinsic pulmonary disease (eg chronic lung disease, or ARDS) as defined by need for positive pressure ventilation, except in association with acute heart failure as determined by the principal investigator
10. Moderate or severe aortic and/or pulmonary valve insufficiency considered technically challenging to repair at the time of the device implantation as determined by the principal investigator
11. Apical VSD or other hemodynamically-significant lesion considered technically challenging to repair at the time of device implantation as determined by the principal investigator
12. Documented heparin induced thrombocytopenia (HIT) or idiopathic thrombocytopenia purpura (ITP) or other contraindication to anticoagulant/antiplatelet therapy
13. Documented coagulopathy (e.g. Factor VIII deficiency, disseminated intravascular coagulation) or thrombophilic disorder (e.g. Factor V Leiden mutation)
14. Hematologic disorder causing fragility of blood cells or hemolysis (e.g. sickle cell disease)
15. Platelets < 70,000/ml within 24 hours prior to device implantation
16. Active infection within 48 hours of implant (positive blood culture OR temperature > 38 degrees C AND wbc > 15,000/ml)
17. Documented human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)
18. Evidence of recent or life-limiting malignant disease
19. Stroke within past 30 days prior to enrollment, or congenital CNS malformation syndrome associated with increased risk of bleeding (e.g. arteriovenous malformation, moya moya)
20. Psychiatric or behavioral disease (e.g. antisocial disorder) with a high likelihood for non-adherence to the protocol and follow-up
21. Currently participating in another investigational device or drug trial and has not completed the required follow-up period for that study. EXCEPTION: Dual enrollment in PUMPKIN study is permitted.
22. Patient is pregnant or nursing

    -

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Number of major bleeding adverse events reported using the Stanford Anti-Thrombotic Protocol. | Up to 90 days
  To test the safety of the Stanford Anti-Thrombotic Protocol.
Number of all forms of stroke events reported using the Stanford Anti-Thrombotic Protocol. | Up 90 days
  To test the effectiveness of the Stanford Anti-Thrombotic protocol.

IPD SHARING:
Plan to Share IPD: No